CLINICAL TRIAL: NCT00457405
Title: Does a Seven Day Treatment With Dipyridamole Induce Protection Against Ischemia-Reperfusion Injury?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: G Rongen, dept Pharmacology Toxicology
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dipy003
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Ischemia-Reperfusion Injury; Atherosclerosis
Keywords: ischemia-reperfusion injury; atherosclerosis; dipyridamole; annexin A5 targeting
MeSH Terms: conditions — Reperfusion Injury; Atherosclerosis | interventions — Dipyridamole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): first 7 day treatment with dipyridamol and at least two weeks later 7 day treatment with placebo
  Interventions: Drug: dipyridamole
- 2 (Active Comparator): first 7 day treatment with placebo and at least two weeks later 7 day treatment with atorvastatin
  Interventions: Drug: dipyridamole

INTERVENTIONS:
Drug: dipyridamole — dipyridamole 200mg twice daily
  Other Names: persantin

SUMMARY:
This study is performed to determine whether a seven day treatment with dipyridamole (slow release, 200mg twice daily) can induce a protective effect against ischemia-reperfusion injury, after ischemic exercise of the non-dominant forearm in healthy volunteers.

DETAILED DESCRIPTION:
Rationale:

Dipyridamole increases the endogenous adenosine level by inhibition of the nucleoside transporter (ENT-1). Activation of the adenosine receptor protects against ischemia-reperfusion injury (pharmacologic preconditioning).

The purpose of this project is to explore whether a seven day treatment with dipyridamole can reduce ischemia-reperfusion injury in the forearm, in a randomized double blind placebo controlled trial.

Study design:

Randomized double-blind placebo-controlled trial with a cross-over design.

Study population:

Healthy male volunteers, aged 18-50 yr

Intervention:

10 Volunteers will be randomised to receive in a cross-over design either a 7 day treatment with dipyridamole (Persantin retard; 200 mg twice daily) or placebo followed by 10 minutes of ischemic isometric muscle contraction of the non-dominant forearm and upon reperfusion infusion of radiolabeled Annexin A5 (Annexin scintigraphy).

Main study parameters/endpoints:

Percentage difference in radioactivity (counts/pixel) between experimental and control thenar muscle at 60 and 240 minutes after reperfusion.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

This study will be executed at the Clinical Research Centre Nijmegen under close medical supervision. Treatment with dipyridamole is not expected to harm the volunteers. During the first days of treatment with dipyridamole, a headache may occur. Ischemic hand gripping will temporarily result in pain in the forearm. This is completely reversible upon reperfusion. Administration of radiolabeled Annexin A5 results in an effective dose of less than 5 mSv, well within the range of accepted exposure to radioactivity for human research. Participation in this research does not interfere with possible diagnostic or therapeutic procedures with X-rays of radioactivity in the future.

Occurrence of an allergic reaction is theoretically possible upon administration of Annexin A5, however there have been no allergic reactions reported in all volunteers exposed to Annexin A5.

The volunteers will not benefit directly from participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male
* age between 18-50yr.

Exclusion Criteria:

* cardiovascular disease
* hypertension (systole > 140 mmHg, diastole > 90 mmHg)
* hypercholesterolemia (fasting total cholesterol > 5.5 mmol/l or not fasting total cholesterol > 6.5mmol/L)
* diabetes mellitus (fasting glucose > 7.0 mmol/L or random glucose > 11.0 mmol/L)
* asthma (recurrent episodes of dyspnea and wheezing, or usage of prescribed inhalation medication: i.e. corticosteroids or B2-agonists)
* participation in any clinical trial during the last 60 days prior to this study.
* administration of any radioactivity for research purposes during the last 5 years prior to this study.
* concomitant medication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Percentage difference in radioactivity (counts/pixel) between experimental and control thenar muscle at 60 and 240 minutes after reperfusion. | 60 and 240 minutes after reperfusion

SECONDARY OUTCOMES:
Plasma dipyridamole concentration | in the morning of day seven of treatment
Workload (duration of exercise and developed force) | during 10 minutes ischemic exercise
Heart rate (preceded by a 7day treatment of dipyridamol or placebo) | during 30 minutes at day seven of treatment with dipyridamol and placebo

CONTACTS AND LOCATIONS:
Overall Officials: G Rongen, MD PhD, Principal Investigator — RUNMC
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Riksen NP, Oyen WJ, Ramakers BP, Van den Broek PH, Engbersen R, Boerman OC, Smits P, Rongen GA. Oral therapy with dipyridamole limits ischemia-reperfusion injury in humans. Clin Pharmacol Ther. 2005 Jul;78(1):52-9. doi: 10.1016/j.clpt.2005.03.003. PMID 16003293